CLINICAL TRIAL: NCT03375840
Title: Pictorial Warning Labels and Memory for Cigarette Health-risk Information Over Time
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Ellen Peters, Professor, Ohio State University
Allocation: Randomized | Model: Factorial | Purpose: Prevention
Other Study IDs: P50CA180908A1; P50CA180908 (NIH)
Record Dates: First submitted 2017-12-08; First posted 2017-12-18 (Actual); Last update posted 2017-12-18 (Actual); Status verified 2017-12

CONDITIONS: Smoking Cessation; Smoking, Cigarette
Keywords: pictorial warning labels; risk knowledge; emotion; memory; risk perceptions; quit intentions
MeSH Terms: conditions — Smoking Cessation; Cigarette Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Text-only PWL, immediate post (Experimental): Exposure to 9 FDA-mandated warning labels
  Posttest measures (e.g., memory, risk perceptions, quit intentions) administered immediately following last exposure to warning labels
  Interventions: Behavioral: Text-only PWL; Behavioral: Immediate posttest
- Text-only PWL, delay posttest (Experimental): Exposure to 9 FDA-mandated warning labels
  Posttest measures (e.g., memory, risk perceptions, quit intentions) administered 6 weeks after last exposure to warning labels
  Interventions: Behavioral: Text-only PWL; Behavioral: delay posttest
- Low-emot PWL, immediate posttest (Experimental): Exposure to 9 warning labels paired with image that elicited little emotion
  Posttest measures (e.g., memory, risk perceptions, quit intentions) administered immediately following last exposure to warning labels
  Interventions: Behavioral: Low-emot PWL; Behavioral: Immediate posttest
- Low-emot PWL, delay posttest (Experimental): Exposure to 9 warning labels paired with image that elicited little emotion
  Posttest measures (e.g., memory, risk perceptions, quit intentions) administered 6 weeks after last exposure to warning labels
  Interventions: Behavioral: Low-emot PWL; Behavioral: delay posttest
- High-emot PWL, immediate posttest (Experimental): Exposure to 9 warning labels paired with image that elicited high emotion
  Posttest measures (e.g., memory, risk perceptions, quit intentions) administered immediately following last exposure to warning labels
  Interventions: Behavioral: High-emot PWL; Behavioral: Immediate posttest
- High-emot PWL, delay posttest (Experimental): Exposure to 9 warning labels paired with image that elicited high emotion
  Posttest measures (e.g., memory, risk perceptions, quit intentions) administered 6 weeks after last exposure to warning labels
  Interventions: Behavioral: High-emot PWL; Behavioral: delay posttest

INTERVENTIONS:
Behavioral: Text-only PWL — Control condition
  Arms: Text-only PWL, delay posttest; Text-only PWL, immediate post
Behavioral: Low-emot PWL — Pictorial warning
  Arms: Low-emot PWL, delay posttest; Low-emot PWL, immediate posttest
Behavioral: High-emot PWL — Pictorial warning
  Arms: High-emot PWL, delay posttest; High-emot PWL, immediate posttest
Behavioral: Immediate posttest
  Arms: High-emot PWL, immediate posttest; Low-emot PWL, immediate posttest; Text-only PWL, immediate post
Behavioral: delay posttest
  Arms: High-emot PWL, delay posttest; Low-emot PWL, delay posttest; Text-only PWL, delay posttest

SUMMARY:
Pictorial cigarette warning labels (PWLs) are thought to increase risk knowledge, but experimental research has not examined PWLs' longer term effects on memory for health risks. This trial tests memory for health risks immediately or after a six-week delay for US-representative adult smokers, US-representative teen smokers/vulnerable smokers, and Appalachian-representative adult smokers. In addition, the trial tests the effects of different warning label components and the consequences of memory for labels on risk perceptions and quit intentions.

ELIGIBILITY:
Inclusion Criteria:

* 19-65 years old (adult samples)
* have smoked 100+ lifetime cigarettes (adult samples)
* currently smoke "every day" or "some days." (adult samples)
* 14-18 years old (teen sample)
* have ever smoked a cigarette (teen sample)

Exclusion Criteria:

• have not ever smoked a cigarette (all samples)

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 4424 (Actual)
Dates: Start 2015-04-17 (Actual); Primary Completion 2016-01-27 (Actual); Study Completion 2016-01-27 (Actual)

PRIMARY OUTCOMES:
graphic warning label recall | immediately following last exposure or after 6-week delay
  free recall for risk information presented in labels (9 text boxes, 1 for each label; coded for exact or equivalent words)
smoking risk recognition | immediately following last exposure or after 6-week delay
  Participants were subsequently shown twenty-six negative health effects and asked "Which of the following health effects were mentioned in the warnings we showed you?" and responded "Yes, I saw this health effect" or "No, I did not see this health effect." Fourteen risks were mentioned in the warnings (e.g., cancer, harms children, emphysema); six were risks of smoking not presented in the warnings (e.g., wrinkles, diabetes), and six were not risks of smoking (e.g., acne, thyroid problems).

SECONDARY OUTCOMES:
smoking risk perceptions | immediately following last exposure or after 6-week delay
  participants completed several scale items about how much risk they perceived smoking posed to them (e.g., "Compared to the average nonsmoker your age, gender, and race, how would you rate your chances of": 1) "getting a life threatening illness because of smoking," 2) "getting lung cancer," and 3) "dying at a younger age than average" (-3 = Much lower, +3 = Much higher))
quit intentions | immediately following last exposure or after 6-week delay
  participants' intentions to quit smoking

REFERENCES:
- [Derived] Peters E, Shoots-Reinhard B, Evans AT, Shoben A, Klein E, Tompkins MK, Romer D, Tusler M. Pictorial Warning Labels and Memory for Cigarette Health-risk Information Over Time. Ann Behav Med. 2019 Mar 20;53(4):358-371. doi: 10.1093/abm/kay050. PMID 29947729